CLINICAL TRIAL: NCT02641496
Title: Cognitive Behavioral Therapy to Increase CPAP Adherence in Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: D1799-R
Record Dates: First submitted 2015-12-22; First posted 2015-12-29 (Estimated); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea; PTSD; Posttraumatic Stress Disorder
Keywords: Obstructive Sleep Apnea; PTSD; Posttraumatic Stress Disorder; Cognitive Behavioral Therapy; Continuous Positive Airway Pressure; CPAP; Cognition; Memory; Quality of Life; Self Efficacy; CBT; OSA; Sleep Apnea; Education; Psychotherapy; Post Traumatic Stress Disorder; Post-Traumatic Stress Disorder; Therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Stress Disorders, Post-Traumatic; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Outcomes Assessor will be masked so as to not influence the 12 month outcome variables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-OSA (Experimental): CBT-OSA is a new cognitive behavioral therapy which focuses on changing behaviors and thoughts to help individuals adjust to using a CPAP machine.
  Interventions: Behavioral: CBT-OSA
- Sleep Education (Active Comparator): The Sleep Education treatment will include information, facts, and videos on sleep, cardiovascular disease, PTSD, and proper sleep hygiene.
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: CBT-OSA — CBT-OSA is a new cognitive behavioral therapy which focuses on changing behaviors and thoughts to help individuals adjust to using a CPAP machine.
  Arms: CBT-OSA
Behavioral: Sleep Education — The Sleep Education treatment will include information, facts, and videos on sleep, cardiovascular disease, PTSD, and proper sleep hygiene.
  Arms: Sleep Education

SUMMARY:
Approximately 20 million Americans suffer from Obstructive Sleep Apnea (OSA) creating risks for major health problems, including dementia, heart attack, and stroke. Obesity, a growing problem for Americans and Veterans alike, is the greatest risk factor for the development of OSA. Male gender and smoking, other OSA risk factors, are common in Veterans. Given the high comorbidity of these risk factors in Veterans, OSA presents a significant health burden to Veterans. The investigators' prior work provides evidence that OSA occurs in up to 69% of Vietnam-era Veterans with Posttraumatic Stress Disorder (PTSD). OSA is easily treated; however, 15-30% of OSA patients are non-compliant with continuous positive airway pressure (CPAP), the standard OSA treatment. The proposed research aims to facilitate adherence to CPAP treatment by testing a novel cognitive-behavioral therapy intervention in Veterans with PTSD. If successful, it may represent an approach that could be applied to the rehabilitation of other chronic conditions with similar barriers to care.

DETAILED DESCRIPTION:
GOALS AND EXPECTED OUTCOMES OF THE PROPOSED RESEARCH The purpose of this proposal is to test a novel cognitive-behavioral therapy (CBT) intervention to increase continuous positive airway pressure (CPAP) treatment adherence for PTSD Veterans with a diagnosis of obstructive sleep apnea (OSA). PTSD is a common, debilitating psychiatric consequence of exposure to trauma and a source of significant disability among U.S. war Veterans. The largest epidemiologic study of PTSD in Vietnam Veterans estimates that 15% of Vietnam Veterans suffer from PTSD [3]. The investigators' research on OSA in Vietnam era Veterans found that 69% of the Veterans in the sample had an Apnea-Hypopnea Index (AHI) 10 [4]. OSA is likely present in 50% of middle-aged and older VA patients [4, 5]. The recurrent hypoxemia and sleep fragmentation associated with OSA can lead to neural injury and functional impairment. Efficacious treatments are available for OSA (e.g., CPAP); however, Veterans with OSA frequently fail to use them [4, 6, 7], leaving these Veterans at risk for cognitive dysfunction [8], deterioration of physical health [9], and negative functional outcomes [10]. The investigators' long-term goal is to improve Veterans' functional outcomes by improving adherence to CPAP. If this intervention proves successful, it may represent an approach that could be applied to the rehabilitation of other chronic conditions with similar barriers to care.

RESEARCH DESIGN AND STRATEGY The reasons for low CPAP adherence include barriers related to discomfort in using CPAP and psychological barriers to behavior change [11]. A CBT treatment to improve CPAP adherence, CBT-OSA, has been successfully applied in civilian randomized controlled trials (RCTs) [12, 13]. The proposed VA intervention would involve delivery of CBT-OSA to PTSD Veterans to foster long-term CPAP adherence. The CBT-OSA treatment would build on the Veterans Integrated Services Network 21 (VISN) Mental Illness Research, Education and Clinical Center's (MIRECC) expertise in CBT interventions [e.g., VA rollout of CBT-Insomnia] as well as on the investigators' current research on PTSD Veterans with OSA. In this sample, the vast majority were not diagnosed with OSA prior to study entry; however, 69% of the participants had an Apnea-Hypopnea Index (AHI) 10 [4]. Of the Veterans previously diagnosed with OSA, 63% were not using their CPAP. Thus, CPAP adherence treatment for PTSD Veterans is the next logical step in the investigators' research. Specifically, the investigators propose a 1-year parallel-group RCT involving 120 PTSD Veterans with a diagnosis of OSA. All participants will receive treatment as usual in VA Pulmonary Service. Participants in the active arm will receive CBT-OSA from a trained Clinical Psychologist. The other arm will receive individual Education based treatment, but not CBT-OSA. Participants in both arms will receive weekly, individual sessions during the first 4 weeks of CPAP treatment and 4 booster sessions during the 1-year protocol. These two arms will be referred to hereafter as the CBT-OSA and the Education groups.

*The investigators will add telehealth treatment as an option for participants due to the COVID-19 pandemic. Research visits may be conducted either in-person or via telehealth (e.g., via video or telephone). Telehealth sessions are subject to approval by the research team. Videoconferencing in particular, requires certain features such as hardware, internet accessibility, and telephone capability.

HYPOTHESES

Hypothesis 1. (Primary) Effect of CBT on CPAP usage. The investigators hypothesize that the CBT-OSA group will use CPAP more hours per night on average than the Education group. ANCOVA will be used to test group differences over time in hours of "mask-on" CPAP usage per night. [Primary endpoint: mean of Days 335-365.]

Hypothesis 2. (Secondary) Effect of CBT on Self-reported Everyday Activities, Mood and Quality of Life. The investigators hypothesize that after initiating CPAP treatment, Veterans in the CBT-OSA group will report more improvement in the ease of performing everyday activities compared to that reported by those in the Education group. ANCOVA will be used to test group differences over time in the total score on the Functional Outcomes of Sleep Questionnaire (FOSQ; [14], at Days 0, 21, 365 (endpoint).

Hypothesis 3. (Secondary) Effect of CBT on Cognitive Outcomes. The investigators hypothesize that the CBT-OSA group will have better cognitive outcomes than the Education group over time. ANCOVA will be applied to the Rey Auditory Verbal Learning Test, Delayed Recall Score with the primary endpoint at Day 365.

Hypothesis 4. (Secondary) Effect of CBT on PTSD. The investigators hypothesize that the CBT-OSA group will have fewer PTSD symptoms than the Education group over time. ANCOVA will be used to test group differences over time in the total score on the PTSD Checklist for DSM-5 (PCL-5), measured at Days 0, 21, 365. Primary endpoint is Day 365.

HOW THE PROPOSED WORK WILL ADDRESS LONGER-TERM GOALS This research fits the VA's goal to reduce functional disabilities in PTSD Veterans with chronic medical conditions. It is designed to not only determine the benefit of this intervention overall, but also to determine in which Veterans CBT-OSA works best. The dataset collected will enable researchers to troubleshoot the intervention and propose improved interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Veterans of any racial or ethnic group
* Age 18 years old and older
* OSA diagnosis by a board-certified Sleep Medicine physician
* Have PTSD
* Capable of giving informed consent for the study; able to read and write English; willing and able to comply with study requirements and restrictions
* Not have a cognitive disorder
* Sufficient visual and auditory acuity for cognitive testing
* No new medication(s) within the prior 1 month. If on a non-excluded medication for a non-excluded condition, the medication regimen will be stable (no changes in dose) for at least 1 month prior to baseline (including anti-hypertensive and diabetic medications).

Exclusion Criteria:

Sleep

* Current CPAP usage, home oxygen therapy, tracheotomy or past corrective surgery for OSA (e.g., uvulopalatopharyngo-plasty, midline glossectomy, or lingualplasty).
* Diagnosis of Central Sleep Apnea (CSA)
* Comorbid sleep disorder
* Working night, rotating or split [period of work, followed by break, and then return to work]; shift work within 1-month of screening or plan to work these shifts during study; Occupations where participants regularly experience jet lag or have irregular work schedules.

Other Medical

* Unstable or moderate to severe chronic illness including systolic congestive heart failure, uncontrolled asthma, severe liver disease, end stage renal disease requiring hemodialysis or history of systemic illness affecting central nervous system (CNS) function (e.g. liver failure, kidney failure, congestive heart failure, systemic cancer).
* Any current clinically significant cardiovascular, respiratory, neurologic, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction unless currently controlled and stable. Any solid organ transplantation.
* Known or suspected neuromuscular disease (e.g. amyotrophic lateral sclerosis, spinal cord injury)
* History of head injury within past year, or history of loss of consciousness > 24 hours
* History of other neurological disease
* Certain medications
* Judged by the investigators to be unable or unlikely to follow the study protocol.

Psychiatric

* Primary psychotic disorder
* Bipolar disorder
* Prominent suicidal or homicidal ideation
* Current exposure to trauma, or exposure to trauma in the past 3 months
* Some substance use
* Presence of acute or unstable psychiatric condition(s) that requires referral for treatment.
* Current or expected cognitive behavior therapy for another condition (e.g. insomnia, anxiety).

Other

* A clinical history or participation in other research that would interfere with the objectives of this study.
* Any other medical, social, or geographical factor that would make it unlikely that the participant would comply with the study procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. Kinoshita, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 133 participants were recruited and screened; 76 met screening requirements, had a working PAP, and completed at least one treatment. From 2019 until study-end, the study was impacted by the departure of Chief Respiratory Therapist, change in study staff, the COVID-19 pandemic (VA halt of PAP distribution and sleep diagnostics from March 2020 to July 2020), national shortage of PAP devices resulting in PAP rationing, and Phillips PAP recall.
Groups:
- CBT-OSA: CBT-OSA is a new cognitive behavioral therapy which focuses on changing behaviors and thoughts to help individuals adjust to using a positive airway pressure (PAP) machine.
  CBT-OSA: CBT-OSA is a new cognitive behavioral therapy which focuses on changing behaviors and thoughts to help individuals adjust to using a PAP machine.
Period: Overall Study
Arm/Group | CBT-OSA | Sleep Education
Started | 41 | 35
Completed | 27 | 23
Not Completed | 14 | 12
Not completed — Lost to Follow-up | 13 | 12
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-OSA | Sleep Education | Total
Number analyzed (Participants) | 41 | 35 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.24 (14.9) | 56.77 (12.11) | 57.03 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 37 | 32 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 31 | 25 | 56
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 3 | 2 | 5
  White | 24 | 20 | 44
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 35 | 76

OUTCOME MEASURES:

1. Primary Outcome: Time in Minutes of "mask-on" Positive Airway Pressure (PAP) Machine Usage Per Night
Description: The PAP machine will measure average PAP use in minutes at two timepoints: first 30 days (encompassing the first four weekly treatment sessions) and the last 30 days (final 30 days of the year long study).
Time Frame: Treatment 1 to Treatment 4 (approximately first 30 days of treatment) and Last 30 Days of 1 Year Study
Population: Of the 50 participants who completed the study, a certain number were missing data for each outcome measure. Only complete data-points were used in the resulting analyses, such that the overall n for mask-on time reflects the total number of participants who had complete data for this particular variable (n=49).
Measure: Mean (Standard Deviation); unit: minutes per night
Groups:
- CBT-OSA: CBT-OSA is a new cognitive behavioral therapy which focuses on changing behaviors and thoughts to help individuals adjust to using a PAP machine.
  CBT-OSA: CBT-OSA is a new cognitive behavioral therapy which focuses on changing behaviors and thoughts to help individuals adjust to using a PAP machine.
Arm/Group | CBT-OSA | Sleep Education
Number analyzed (Participants) | 26 | 23
minutes per night
  Average PAP Use for First 30 Days | 234.00 (140.01) | 144.25 (159.97)
  Average PAP Use for Last 30 Days | 157.04 (161.82) | 152.39 (157.36)
Statistical Analysis 1: Comparison: CBT-OSA vs Sleep Education; Treatment 1 to Treatment 4 (approximately first 30 days of treatment); Test type: Other — ANOVA; p = 0.027, ANOVA — Significance threshold p<0.05; one-tailed
Statistical Analysis 2: Comparison: CBT-OSA vs Sleep Education; Last 30 Days of 1 Year Study; Test type: Other — ANOVA; p = 0.919, ANOVA — Significance threshold p<0.05; one-tailed

2. Secondary Outcome: Functional Outcomes of Sleep Questionnaire (FOSQ)
Description: Effect of CBT on Self-reported Everyday Activities, Mood and Quality of Life. Functional Outcomes of Sleep Questionnaire (FOSQ) total scores range from 5 to 20. Lower values indicate higher functioning across different functional areas (e.g., less interference of fatigue on work functioning or on relationships).
  The investigators hypothesize that after initiating CPAP treatment, Veterans in the CBT-OSA group will report more improvement in the ease of performing everyday activities compared to that reported by those in the Education group.
Time Frame: 1 year
Population: Of the 50 participants who completed the study, a certain number were missing data for each outcome measure. Only complete data-points were used in the resulting analyses, such that the resulting n for FOSQ reflects the total of participants who had complete data for this particular variable (n=40).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-OSA | Sleep Education
Number analyzed (Participants) | 22 | 18
score on a scale | 15.77 (4.03) | 15.10 (3.31)
Statistical Analysis 1: Comparison: CBT-OSA vs Sleep Education; Test type: Other; p = 0.696, ANOVA — Significance threshold p<0.05; one-tailed

3. Secondary Outcome: California Verbal Learning Test, Second Edition (CVLT-II)
Description: Effect of CBT on Cognitive Outcomes. California Verbal Learning Test-II Long Delay Free Recall (CVLT-II LD FC) scores range from 0 to 16. Higher raw scores indicate more items retained and better memory performance.
  The investigators hypothesize that after initiating CPAP treatment, the CBT-OSA group will have better cognitive outcomes than the Education group over time. The California Verbal Learning Test-II, Delayed Recall Score is the cognitive outcome measure.
Time Frame: 1 year
Population: Of the 50 participants who completed the study, a certain number were missing data for each outcome measure. Only complete data-points were used in the resulting analyses, such that the resulting n for CVLT-II Long Delay reflects the total of participants who had complete data for this particular variable (n=45).
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | CBT-OSA | Sleep Education
Number analyzed (Participants) | 24 | 21
raw score | 9.00 (3.16) | 8.48 (3.36)
Statistical Analysis 1: Comparison: CBT-OSA vs Sleep Education; Test type: Other; p = 0.593, ANOVA — Significance threshold p<0.05; two-tailed

4. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: Effect of CBT on PTSD. PTSD Checklist for DSM-5 (PCL-5) total scores range from 0 to 80. For the PCL-5, higher values indicate higher levels of current PTSD symptoms, thus a higher level of current PTSD severity.
  The investigators hypothesize that after initiating CPAP treatment, the CBT-OSA group will have fewer PTSD symptoms than the Education group over time. The PTSD Checklist for DSM-5 (PCL-5) will be the PTSD outcome measure.
Time Frame: 1 year
Population: Of the 50 participants who completed the study, a certain number were missing data for each outcome measure. Only complete data-points were used in the resulting analyses, such that the resulting n for PCL-5 reflects the total of participants who had complete data for this particular variable (n=48).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-OSA | Sleep Education
Number analyzed (Participants) | 26 | 22
score on a scale | 27.31 (18.31) | 26.82 (17.39)
Statistical Analysis 1: Comparison: CBT-OSA vs Sleep Education; Test type: Other; p = 0.925, ANOVA — Significance threshold p<0.05; one-tailed

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected from the time of study entry until end of study participation for each participant, spanning approximately 12 months.
Arm/Group | CBT-OSA | Sleep Education
All-Cause Mortality (participants affected / at risk) | 2/41 | 1/35
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/35
Other Adverse Events (participants affected / at risk) | 5/41 | 1/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-OSA (N=41) | Sleep Education (N=35)
Renal Infarct (Renal and urinary disorders) | 0 (0) | 1 (1) — Renal infarct
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0) — Right-sided cerebrovascular accident
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-OSA (N=41) | Sleep Education (N=35)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Surgery (Surgical and medical procedures) | 4 (4) | 0 (0)
Psychological Distress (Social circumstances) | 1 (1) | 0 (0) — Participant's home burned down in wildfires.

LIMITATIONS AND CAVEATS:
Participant recruitment was impacted heavily throughout the study for various reasons. From 2019 until study-end, the study was impacted by the departure of Chief Respiratory Therapist, change in study staff, the COVID-19 pandemic (VA halt of PAP distribution and sleep diagnostic testing from March 2020 to July 2020), Phillips PAP recall, and national shortage of PAPs (significant PAP rationing: PAPs only prescribed to patients at imminent risk of death/hospitalization without PAP therapy).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT02641496/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT02641496/SAP_001.pdf
  • Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT02641496/ICF_002.pdf